CLINICAL TRIAL: NCT00412308
Title: A Comparison of High vs. Low Tidal Volumes in Ventilator Weaning for Individuals With Sub-Acute Cervical Spinal Cord Injuries
Brief Title: A Comparison of High vs. Low Tidal Volumes in Ventilator Weaning for Individuals With Cervical Spinal Cord Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Craig Hospital (Other)
Responsible Party: Daniel Lammertse, MD, Craig Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H133N060005
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Spinal Cord Injury; Respiratory Insufficiency
Keywords: spinal cord injury; ventilator dependency; ventilator weaning; tidal volume
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Insufficiency | interventions — Respiration, Artificial

INTERVENTIONS:
Procedure: Tidal volume used in mechanical ventilation

SUMMARY:
The study will compare outcomes between individuals with sub-acute, ventilator-dependent tetraplegia using high (20 cc/kg) vs. low (10 cc/kg) tidal volumes during mechanical ventilator support.

DETAILED DESCRIPTION:
While respiratory failure in people with SCI is common, clinicians have not come to a consensus on the best strategy to manage the mechanical ventilation of these individuals or whether to manage people with SCI differently from other patients. The Consortium for Spinal Cord Medicine has developed Clinical Practice Guidelines using protocols established at Craig Hospital in the 1980s and 1990s, but these are based only on clinical experience and retrospective, cohort data using historical controls.

These guidelines suggest that patients should be ventilated with tidal volumes (VT)of 20-25 cc/kg of ideal body weight (IBW). This recommended VT is at least twice as large as conventional VT used for general medical and surgical patients requiring mechanical ventilation. However, there is a clinical belief that people with SCI should be ventilated at higher VT to prevent atelectasis, to decrease the risk of pneumonia, and to facilitate weaning. This belief was fostered by a retrospective, concurrent cohort comparison study of individuals with SCI, which found that the use of high VT on the ventilator (mean 25.3 cc/kg, PAP<40) was associated with more rapid resolution of atelectasis and more rapid weaning from mechanical ventilation than the use of low VT (mean 15.5). Therefore, people with SCI have been clinically managed using high VT for the past 2-3 decades without prospective data to confirm these clinical impressions.

At the same time that these ventilator strategies evolved in the care of patients with SCI, several clinical studies in general medical and surgical patients requiring mechanical ventilation suggested that high VT leading to higher airway pressures could actually promote lung injury. This occurred when higher VT increased the risk of over-distending the airways and creating volume-related trauma.16-19 In multiple studies, VT of only 10-15 cc/kg IBW was found to produce alveolar over-distention, stretch injury and barotrauma. This work led to the belief that low VT of 6-8 cc/kg IBW could be helpful in protecting mechanically ventilated individuals from ventilator-induced lung injury.

Whether these findings and recommendations apply to individuals with SCI requiring mechanical ventilation is unclear. At least one study of mechanically ventilated individuals without acute respiratory distress syndrome suggests that the use of low VT (6 cc/kg) increases the risk of atelectasis.

With the lack of prospective, evidence-based data regarding optimal VT for persons with a SCI who are ventilator-dependent, clinicians may be inclined to use lower VT to prevent lung injury, unless there is more definitive data to show that higher volumes are as safe as low VT and that higher VT facilitate more rapid weaning from mechanical ventilation.

This is a prospective randomized, controlled study to compare outcomes between individuals with sub-acute, ventilator-dependent tetraplegia using high (20 cc/kg) tidal volume (VT) vs. low (10 cc/kg) VT during mechanical ventilator support. While the use of lower tidal volumes in the general pulmonary community is more common, we and others in the SCI rehabilitation community have used 20 cc/kg IBW tidal volumes or higher to manage and attempt to wean individuals with SCI on mechanical ventilation. This study will address the safety and efficacy of using higher VT in ventilator weaning. A series of objective measures and standardized protocols are implemented to ensure equivalent pulmonary management and weaning processes in individuals, regardless of their randomization status.

* For individuals with sub-acute ventilator-dependent tetraplegia, providing high tidal volumes (VT = 20 cc/kg) will result in more rapid weaning from mechanical ventilation than use of low tidal volumes (VT = 10 cc/kg) in an 8-week trial.
* For these individuals, use of high tidal volumes will result in fewer episodes of atelectasis and ventilator acquired pneumonia (VAP) compared to use of low tidal volumes.
* There will be no difference in the incidence of a) barotrauma or b) ARDS between those using high tidal volumes compared to those using low tidal volumes.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI at levels C3 through C6, ASIA A, B, or C tetraplegia
* Subacute admission to Craig Hospital between 2 weeks and 6 months post-injury
* Completely ventilator-dependent (24 hours a day) at the time of admission to Craig Hospital
* Age 18-55 years
* Informed consent obtained

Exclusion Criteria:

* Concurrent severe traumatic brain injury resulting in inability to cooperate with wean protocol
* Residual severe chest trauma (pneumothorax, recurrent pleural effusion > one third hemithorax, indwelling chest tubes, flail chest, trapped lung, bilateral pulmonary contusions)
* Residual esophageal trauma that may cause ongoing aspiration;
* Current ARDS
* Current VAP unresponsive to antibiotic therapy
* Premorbid cardiomyopathy with ejection fraction <30%, unstable angina, bullous emphysema, obstructive lung disease with forced expiratory volume < 50% predicted, morbid obesity with BMI ≥ 35, increased intracranial pressure, neuromuscular disease, chronic liver disease Child-Pugh Class C, or history of bone marrow or solid organ transplantation
* Critical illness polyneuropathy
* Burns over more than 30 percent of their body-surface area
* Current participation in another clinical trial
* Any condition that, in the judgment of the investigator, precludes successful participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-12; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Time to full weaning from ventilator
Episodes of atelectasis
Episodes of ventilator-acquired pneumonia
Episodes of barotrauma
Episodes of acute respiratory distress syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Mary Warner, MD, Principal Investigator — South Denver Pulmonary Associates PC; James Fenton, MD, Principal Investigator — South Denver Pulmonary Associates, PC; Daniel P Lammertse, MD, Principal Investigator — Craig Hospital
Locations (1):
- Craig Hospital, Englewood, Colorado, United States